CLINICAL TRIAL: NCT07249593
Title: Parental Recognition of Child Needs and Its Impact on Early Childhood Regulatory Problems
Brief Title: Recognizing Children's Needs: Impact on Early Childhood Regulatory Problems
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Division of Social Pediatrics, Marmara University School of Medicine, Marmara University
Other Study IDs: 27.05.2025-46
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Regulation, Self; Reflective Functioning; Mentalization; Child Sleep; Parent-Child Relation; Crying; Feeding Problems
Keywords: regulatory problems; maternal sensitivity; sleep; feeding; crying; Parental reflective functioning; Mentalization; Insightfulness
MeSH Terms: conditions — Self-Control; Crying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary:

This study aims to quantitatively examine the relationship between regulatory problems (sleep, feeding, and crying) in infants aged 6-36 months and levels of parental sensitivity and reflective functioning. The primary objective is to determine how parents' ability to perceive and interpret their child's cues affects these regulatory difficulties; the secondary objective is to explore how emotional responses to crying and other parent-child interaction factors mediate that relationship. In a cohort of approximately 249 infant-parent dyads, the Revised-Brief Infant Sleep Questionnaire (BISQ-R), feeding and crying assessment forms, the Parental Reflective Functioning Questionnaire, the My Emotions Questionnaire, and the Parental Stress Scale will be administered. Data will be analyzed via descriptive statistics, correlation analyses, and multiple regression models. As the first large-scale quantitative study in Turkey to investigate this area, it will yield unique data to guide parenting programs and early-intervention policies.

DETAILED DESCRIPTION:
Regulatory difficulties in early childhood are commonly manifested as excessive crying in infants over three months old, and as feeding and sleep problems in infants over six months old. These difficulties are prevalent and are believed to be related to later problems with self-regulation. When sleep, feeding, and crying problems are considered together as regulation difficulties, prevalence estimates during the first year of life are approximately 20%, and co-occurrence of more than one regulation problem has been reported in 2-8% of cases. Although many early regulation difficulties are transient, they have been associated with later social and behavioral problems in childhood and with cognitive and behavioral difficulties in adulthood in longitudinal studies. Regulation difficulties are best understood within a transactional model in which infant temperament, caregiver behaviors, parental psychopathology, parental perceptions of infant behaviors, and broader sociocultural and environmental factors interact to shape infant sleep, feeding, and crying patterns. The dynamic relationship between parents and infants plays a critical role in the development of sleep problems. Whether the parent perceives the infant's sleep characteristics as problematic is influenced by many factors, and this, in turn, affects parental behaviors during the infant's nighttime awakenings. As a result, sleep problems are among the early regulation issues and are closely related to parent-child interactions. Parental sensitivity and parental reflective functioning (i.e., the caregiver's capacity to understand both their own and their child's mental states) are key proximal determinants of how regulation difficulties develop and how they are managed. Temperament and regulation difficulties overlap conceptually but are distinct constructs: temperament refers to biologically based individual differences in reactivity and self-regulation that evolve through reciprocal interactions with caregivers. Importantly, the relation between temperament and regulation difficulties is moderated by caregiving behaviors, highlighting the clinical importance of identifying temperament to provide tailored parenting recommendations. Caregiver-infant interaction during early childhood forms the foundation for social, emotional, and cognitive development. Caregiver sensitivity, defined as the ability to notice, accurately interpret, and promptly, consistently, and appropriately respond to infant signals (e.g., crying, smiling, gaze, and movement), is a major contributor to the development of healthy self-regulation. Parental reflective functioning (also referred to as parental mentalization, mind-mindedness, or insightfulness) describes the caregiver's capacity to consider the child's inner mental states and to view events from the child's perspective, and it is closely linked to sensitive caregiving. High caregiver sensitivity and reflective functioning support the child's ability to have their feelings and needs recognized and responded to, which may bolster the development of self-regulatory capacities.This study examines the relationship between caregivers' capacity to understand and interpret their infant's behaviors (i.e., parental reflective functioning and sensitivity) and infants' self-regulatory abilities, operationalized by sleep, feeding, and crying regulation measures. By clarifying these relationships, the research aims to inform interventions that enhance caregiver responsiveness and tailored caregiving strategies to reduce early regulation difficulties and their downstream developmental consequences.The primary aim of this study is to determine the effect of the parent's capacity to understand the infant's behaviors on regulation problems observed during early childhood (6-36 months). The secondary aims are to examine the emotional responses of mothers to infant crying and the mediating role of child and parent-related factors in this relationship. The research aims to contribute to the understanding of regulation problems through variables such as parental behaviors and child temperament characteristics.The study will be conducted through the online surveys, but it will be administered individually by the researcher, targeting the parents of infants in early childhood. This study adopts a longitudinal, prospective design. Mothers who have a 6 months old infant will be invited to participate. Recruitment will take place from December 2025 to March 2026. Mothers will be followed across four time points: 6, 12, 18, and 36 months of the child's age. Sociodemographic information will also be collected. Mothers will be assessed using the Parental Reflective Functioning Questionnaire, Parental Stress Scale, and My Emotions Questionnaire. The sleep of children will be evaluated by the Turkish version of the Revised-Brief Infant Sleep Questionnaire, feeding and crying problems will be assessed using the methodology established by Bilgin A. et al. Child's temperament will be assessed using the Early Childhood Behavior Questionnaire Very Short Form.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older with a infant aged 6 months (± 1 month)
* Willingness to participate in the study and follow-up
* Ability to speak, understand and communicate fluently in Turkish.

Exclusion Criteria:

* Mothers of infants with serious chronic conditions requiring follow-up, diagnosed after birth, even if included in the study
* Individuals who completed the questionnaire but did not meet the questionnaire reliability criteria
* Parents of babies with a history of preterm birth (gestational age under 37 weeks)
* Parents of babies with a history of low birth weight (<2500g)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy mothers aged 18 and above and her healthy children 0-36 months
Sampling Method: Non-Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Infant sleep-wake patterns | 6th, 12th, 18th and 36th months
  Infant sleep-wake patterns will be measured using the Revised-Brief Infant Sleep Questionnaire (BISQ-R). The BISQ-R is a parent-reported screening tool designed to evaluate sleep patterns in infants and young children. This scale consists of 33 questions with 19 questions for scoring. There are 3 subscales including infant sleep, parent perception, and parent behavior. The total and each subscale score ranges from 0 to 100. The total score is the average of the 3 subscale scores. Higher scores indicate better sleep quality, more positive perception of infant sleep, and parental behaviors that promote healthy and independent sleep. The survey has been validated in Turkish.
Infant Crying | 6th, 12th and 18th months
  Crying: In the present study, the assessment of crying will be conducted in accordance with the methodology employed in the research conducted by Bilgin A. et al.. A child will be considered to have a crying problem if at least one of the following three measures is present:
  * At 6 months:
    1. Crying for 120 minutes or more (assessed as Yes/No)
    2. Difficulty or great difficulty soothing the baby (Easy/Difficult)
    3. Mother perceives the crying as disturbing (assessed as Yes/No)
  * At 12 months:
    1. Crying for 60 minutes or more (assessed as Yes/N(note: this data is not available in the Bilgin A.'s study-only collected at 0, 3, 6, and 18 months)o)
    2. Difficulty or great difficulty soothing the baby (Easy/Difficult)
    3. Mother perceives the crying as disturbing (assessed as Yes/No)
  * At 18 months:
    1. Crying for 60 minutes or more (assessed as Yes/No)
    2. Difficulty or great difficulty soothing the baby (Easy/Difficult)
    3. Mother perceives the crying as disturbing (assessed as Yes/No)
Feeding | 6th, 12th and 18th months
  Feeding: In the present study, the feeding will be assessed in accordance with the methodology employed by Bilgin A. et al. Feeding problems will be evaluated in participants using two general items. This section will assess selective eating/food refusal.
  * At 6 months: fighting with breast/bottle will be assessed (Yes/No).
  * At 12 and 18 months: selective eating/food refusal will be assessed by asking the following items (Yes/No for each):
    1. eating very little
    2. leaving most of the food offered
    3. lack of appetite
    4. being selective about foods
    5. eating slowly
    6. refusing lumpy/textured foods
    7. even refusing pureed foods

SECONDARY OUTCOMES:
Parental Reflective Functioning | 6th, 12th, 18th and 36th months
  Parental Reflective Functioning will be measured using the Parental Reflective Functioning Questionnaire (PRFQ). The PRFQ is an 18 item parent report instrument with three subscales: Interest and Curiosity (IC), Certainty about Mental States (CMS), and Pre mentalizing Modes (PM). Items are rated on a 7 point Likert scale (1 = strongly disagree to 7 = strongly agree). Subscale scores reflect distinct aspects of parental mentalizing (IC: interest in the child's mental states; CMS: tolerance of uncertainty about mental states; PM: non mentalizing or maladaptive attributions), and higher scores have different interpretations depending on the subscale. The measure has demonstrated acceptable internal consistency in validation studies and a validated Turkish short form is available.
Mother's Emotional Reactions | 6th, 12th, 18th and 36th months
  My Emotions Questionnaire (MEQ) will be used to assess mothers' emotional responses to infant crying. The MEQ is a 20 item parent report measure comprising five subscales: Amusement, Anxiety, Frustration, Sympathy, and Protective. Items are summed to produce subscale and total scores (range 20-100); higher scores indicate more frequent or problematic emotional responses. A Turkish reliability and validity study of this questionnaire will be conducted concurrently. Permission for use and ethics committee approval has been obtained.
Temperament | 18th and 36th months
  Early Childhood Behavior Questionnaire - Very Short Form (ECBQ VSF) will be administered as a parent report measure of temperament for children aged 18th and 36th months. The ECBQ VSF contains 36 items rated on a 7 point Likert scale (1 = never to 7 = always) and yields three subscale scores: Negative Affectivity, Surgency (Extraversion), and Effortful Control. Each subscale score is calculated as the mean of its constituent item scores (items requiring reverse scoring should be recoded prior to averaging). Higher scores indicate greater expression of the corresponding temperament dimension (e.g., higher Negative Affectivity -more frequent/intense negative emotion; higher Effortful Control = stronger self regulation).
Parental Stress Level | 6th, 12th, 18th and 36th months
  Parenting Stress Scale (PSS) will be used for parent reported measure of parenting stress. The PSS is a 16 item, 5 point Likert scale (1 = strongly disagree to 5 = strongly agree) that assesses perceived stress related to parenting. Total scores range from 16 to 80, with higher scores indicating greater parenting stress. The scale is organized into four subscales: Parental Rewards, Parental Stressors, Lack of Control and Parental Satisfaction. The maximum score is 80, and the minimum score is 16. Higher scores indicate more problematic responses.
Behavior | 18th and 36th months
  Early Childhood Behavior Questionnaire - Very Short Form (ECBQ VSF) will be administered as a parent report measure of temperament for children aged 18th and 36th months (19). The ECBQ VSF contains 36 items rated on a 7 point Likert scale (1 = never to 7 = always) and yields three subscale scores: Negative Affectivity, Surgency (Extraversion), and Effortful Control. Each subscale score is calculated as the mean of its constituent item scores (items requiring reverse scoring should be recoded prior to averaging). Higher scores indicate greater expression of the corresponding temperament dimension (e.g., higher Negative Affectivity -more frequent/intense negative emotion; higher Effortful Control = stronger self regulation).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Requests for wider sharing of data (for example in response to information on Marmara University webpages and in publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate and meets the criteria set by the university; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.

REFERENCES:
- [Background] Gördesli, M. A., & Sünbül, Z. A. (2021). The psychometric properties of parental stress scale-Turkish Form. Turkish Psychological Counseling and Guidance Journal, 11(61), 199-213.
- [Background] Putnam SP, Gartstein MA, Rothbart MK. Measurement of fine-grained aspects of toddler temperament: the early childhood behavior questionnaire. Infant Behav Dev. 2006 Jul;29(3):386-401. doi: 10.1016/j.infbeh.2006.01.004. Epub 2006 Mar 2. PMID 17138293
- [Background] Arikan G, Acar IH, Ustundag-Budak AM. A two-generation study: The transmission of attachment and young adults' depression, anxiety, and social media addiction. Addict Behav. 2022 Jan;124:107109. doi: 10.1016/j.addbeh.2021.107109. Epub 2021 Sep 3. PMID 34547644
- [Background] Baris HE, Us MC, Boran P. Turkish adaptation of the maternal cognition about infant sleep questionnaire. Sleep Med X. 2023 Dec 29;7:100102. doi: 10.1016/j.sleepx.2023.100102. eCollection 2024 Dec. PMID 38268570
- [Background] Grienenberger JF, Kelly K, Slade A. Maternal reflective functioning, mother-infant affective communication, and infant attachment: exploring the link between mental states and observed caregiving behavior in the intergenerational transmission of attachment. Attach Hum Dev. 2005 Sep;7(3):299-311. doi: 10.1080/14616730500245963. PMID 16210241
- [Background] Slade A, Grienenberger J, Bernbach E, Levy D, Locker A. Maternal reflective functioning, attachment, and the transmission gap: a preliminary study. Attach Hum Dev. 2005 Sep;7(3):283-98. doi: 10.1080/14616730500245880. PMID 16210240
- [Background] Meins E, Fernyhough C, Fradley E, Tuckey M. Rethinking maternal sensitivity: mothers' comments on infants' mental processes predict security of attachment at 12 months. J Child Psychol Psychiatry. 2001 Jul;42(5):637-48. PMID 11464968
- [Background] Koren-Karie N, Oppenheim D, Yuval-Adler S, Mor H. Emotion dialogues of foster caregivers with their children: the role of the caregivers, above and beyond child characteristics, in shaping the interactions. Attach Hum Dev. 2013;15(2):175-88. doi: 10.1080/14616734.2013.746822. Epub 2012 Nov 27. PMID 23186141
- [Background] Leerkes EM, Qu J. The My Emotions Questionnaire: A self-report of mothers' emotional responses to infant crying. Infant Ment Health J. 2020 Jan;41(1):94-107. doi: 10.1002/imhj.21830. Epub 2019 Sep 11. PMID 31508839
- [Background] Ainsworth, M. D. S., Blehar, M. C., Waters, E., & Wall, S. N. (2015). Patterns of attachment: A psychological study of the strange situation. Psychology press.
- [Background] Sidor A, Fischer C, Cierpka M. The link between infant regulatory problems, temperament traits, maternal depressive symptoms and children's psychopathological symptoms at age three: a longitudinal study in a German at-risk sample. Child Adolesc Psychiatry Ment Health. 2017 Mar 6;11:10. doi: 10.1186/s13034-017-0148-5. eCollection 2017. PMID 28286548
- [Background] Stuhrmann LY, Gobel A, Bindt C, Mudra S. Parental Reflective Functioning and Its Association With Parenting Behaviors in Infancy and Early Childhood: A Systematic Review. Front Psychol. 2022 Mar 3;13:765312. doi: 10.3389/fpsyg.2022.765312. eCollection 2022. PMID 35310277
- [Background] Leerkes EM. Predictors of Maternal Sensitivity to Infant Distress. Parent Sci Pract. 2010 Jul 1;10(3):219-239. doi: 10.1080/15295190903290840. PMID 20824194
- [Background] Sadeh A, Tikotzky L, Scher A. Parenting and infant sleep. Sleep Med Rev. 2010 Apr;14(2):89-96. doi: 10.1016/j.smrv.2009.05.003. Epub 2009 Jul 23. PMID 19631566
- [Background] Wolke D, Baumann N, Jaekel J, Pyhala R, Heinonen K, Raikkonen K, Sorg C, Bilgin A. The association of early regulatory problems with behavioral problems and cognitive functioning in adulthood: two cohorts in two countries. J Child Psychol Psychiatry. 2023 Jun;64(6):876-885. doi: 10.1111/jcpp.13742. Epub 2023 Jan 5. PMID 36601777
- [Background] Bilgin A, Baumann N, Jaekel J, Breeman LD, Bartmann P, Bauml JG, Avram M, Sorg C, Wolke D. Early Crying, Sleeping, and Feeding Problems and Trajectories of Attention Problems From Childhood to Adulthood. Child Dev. 2020 Jan;91(1):e77-e91. doi: 10.1111/cdev.13155. Epub 2018 Oct 6. PMID 30291757
- [Background] Hemmi MH, Wolke D, Schneider S. Associations between problems with crying, sleeping and/or feeding in infancy and long-term behavioural outcomes in childhood: a meta-analysis. Arch Dis Child. 2011 Jul;96(7):622-9. doi: 10.1136/adc.2010.191312. Epub 2011 Apr 20. PMID 21508059
- [Background] Bilgin A, Wolke D. Regulatory Problems in Very Preterm and Full-Term Infants Over the First 18 Months. J Dev Behav Pediatr. 2016 May;37(4):298-305. doi: 10.1097/DBP.0000000000000297. PMID 27096573